CLINICAL TRIAL: NCT04051918
Title: Robot-Assisted Cognitive Training for Socially Isolated Older Adults With Mild Cognitive Impairment
Brief Title: Robot-assisted Cognitive Training for Lonely Older Adults With Mild Cognitive Impairment (MCI)
Acronym: MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Georgia (Other)
Collaborators: Applied Universal Dynamics, Corp. (Unknown); Van Robotics, Inc. (Unknown)
Responsible Party: Principal Investigator, Jenay M. Beer, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PROJECT00000940
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Cognitive Change; Cognitive Impairment, Mild; Aging
Keywords: cognitive training; socially assistive robotics; music learning
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Older adults with mild cognitive impairment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socially Assistive Robot Intervention (Experimental): Piano training intervention led by a semi-autonomous socially assistive robot
  Interventions: Behavioral: Piano Training
- Content Only Intervention (Active Comparator): Piano training intervention using the same curriculum displayed on a computer monitor, without the socially assistive robot tutor.
  Interventions: Behavioral: Piano Training

INTERVENTIONS:
Behavioral: Piano Training — Cognitive training via music learning

SUMMARY:
This study will use a socially assistive robot to deliver cognitive training in the form of a music (piano) learning intervention to socially isolated older adults with mild cognitive impairment.

DETAILED DESCRIPTION:
Cognitive training has been shown in past research to improve cognitive function in older adults with and without mild cognitive impairment. Music learning has been previously shown to be a particularly effective form of cognitive training: in addition to the cognitive demands of learning notation, hand positioning, coordination and timing, those who engage in music learning also benefit from emotional connection to the music and social engagement with a music teacher.

Not all older adults are able to access music lessons. Older adults who are homebound, live in rural areas and do not have access to reliable transportation (or a monthly income with sufficient funds for recurring payments for lessons) are unlikely to be able to access these benefits. Socially assistive robots that can deliver both education and companionship on an ongoing basis within the home environment may be a viable solution to these limitations.

The purpose of this study is to deliver cognitive training in the form of a music (piano) learning intervention to older adults who are socially isolated, and who may be able to benefit from the cognitive training aspects of the intervention. A socially assistive robot will deliver the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be able to speak, read and write in English with a high degree of fluency
* Cumulative music learning experience < 3 years
* Able to sit upright for two hours at a time
* Able to see images on a screen at a distance of approximately 20 inches
* Must have independent transportation to and from the Institute of Gerontology, weekly, for 27 weeks
* No hearing impairment beyond what is correctable via hearing aid
* Must have a safe location in the home to store and use an 88-key keyboard + stand and piano bench
* No more than mildly cognitively impaired: global deterioration scale no higher than 2-3; Clinical Dementia Rating Scale no higher than 0.5 (sum of boxes)
* Must have a close companion, family member or loved one who can attend the first and last visit
* Must be capable of providing informed consent (based on responses to questions on study purpose, tasks, benefits, incentives and risks).
* Must have a computer or tablet that is connected to broadband internet, to be used three times over the course of the study
* Must have access to an e-mail account that can be checked three times during the study

Exclusion criteria:

* No previous diagnosis of Alzheimer's disease or related dementias
* No condition that limits movement of the hands or fingers

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Verbal Memory Test | 6-months
  Correct hits + Correct passes + Correct hits after 30-minute delay + Correct passes after 30-minute delay; higher score is better; items remembered from a word list that also contains distractors
Visual Memory Test | 6-months
  Correct hits + Correct passes + Correct hits after 30-minute delay + Correct passes after 30-minute delay; higher score is better; images remembered from an image list that also contains distractors
Non-Verbal Reasoning Test | 6-months
  correct responses - commission errors; higher score is better
Shifting Attention Test | 6-months
  correct responses - errors; higher is better
Stroop Test | 6-months
  [Simple RT < (Complex RT Correct *0.1)+Complex RT Correct] AND [Complex RT Correct < ( Stroop RT Correct *0.1)+Stroop RT Correct] AND (Complex Correct > Complex Errors) AND (Stroop Correct > Stroop Errors)
Continuous Performance Test | 6-months
  CPT Correct Responses >= 30 AND CPT Correct Responses > CPT Commission Errors
Symbol Digit Coding Test | 6-months
  SDC Correct Responses >= 20 AND Correct Responses > Errors

SECONDARY OUTCOMES:
Technology Acceptance - TAM3 | 6-months
  higher sore = greater acceptance
DeJong Loneliness Scale | 6-months
  Higher scores indicate more severe loneliness
NASA TLX | 6-months
  Measures workload; higher score = more work

OTHER OUTCOMES:
Global deterioration scale | 6-months
  Staging of cognitive impairment based on a structured clinical interview; higher score = more severe impairment

CONTACTS AND LOCATIONS:
Overall Officials: Jenay Beer, Ph.D., Principal Investigator — The University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with researchers outside of the study site.